Originally developed: 01/01 2023

Does Manual Treatment With Craniosacral Therapy Change the Experience of Dry Mouth in People Who Suffers From Dry Mouth After Cancer in Throat Or Mouth - a Pilot Study

NCT05882890

Participants in the research project have been using a standard informed consent form in Danish made by the Danish Research Ethics Committees

## Consent to publication of the research results from the project

Efficacy of Manual Treatment of Tissue in the Diaphragm, Throat, Neck, Cranium and Mouth Region for Radiation-induced Xerostomia and Hypo- or Subnormal Salivation - a case study

(title is later changed to: Does Craniosacraltherapy Combined With Exercises That Focuses om Respiration and Posture in the Upper Body Have an Effect on Xerostomia and Other Late Sequelae on People Who Has Been Suffering From Cancer in Mouth and Throat?

The results in this project contains personal information about you in pseudo-anonymized form. Therefore it is my duty to obtain your written consent to publish the results from the project.

The purpose of this consent is to obtain your permission for me (Cathrine Rahbek) to publish the results from the research project in oral and written form.

### Which personal health information will be published?

The health information contains, among other things:

- number of years since cancer
- location of tumor and which treatment you received for the cancer
- age
- sex
- what late effects you have after your treatment
- what, if any, effect you have after receiving the treatment in this project

The information is given in the form "10 out of 10 points in experiencing dry mouth"

In addition the results (average from the replies in the questionnaire "dry mouth after at least 3 month") will be published.

The results will be published in a pseudo-anonymized form – that means that your identity can only be found, if the published result is combined with prior knowledge about you. I will of course not publish or give such knowledge to anyone.

#### Where will the the information be published?

The research results will be published in oral form in presentation, and in written form to relevant patient associations and relevant professionals.

I addition I plan to publish the results on "Upledger International's" home page, and maybe the association of craniosacral therapists in Denmark. Maybe the results will also be accessible at the "Association of Danish Physiotherapist's" home page. If possible it will also be published in a scientific journal.

In addition I will refer to it on my webside.

# Withdrawal of your consent

It is my duty to inform you at that you can, at any time, withdraw your consent to puplication of the results. If that happens I will to the extent possible withdraw links and information in written form from all available places where the information is freely available and remove your information BUT if the results has been published in a scientific journal it will not be possible.

## **Voluntarily and informed consent**

| When signing this, you are also stating that your consent is being given voluntarily and on an |
|---|
| informed basis. |
| Signature/date |